CLINICAL TRIAL: NCT01752335
Title: Effect of Monoclonal Anti-IL6 Antibody (Tocilizumab) on the Cardiovascular Risk in Patients With Rheumatoid Arthritis
Acronym: TOCRIVAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FRC-TOC-2009-01; 2010-018658-12 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-19 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, tocilizumab, cardiovascular risk factors
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tocilizumab (Other): All the patients are treated with tocilizumab before inclusion. The doses, frequency and duration are in acordance with the Summary of Characteristics of the Product authorised by EMA.
  Usually 8mg/kg (not minor than 480 mg), once each 4 weeks.
  Interventions: Other: Braquial ecography

INTERVENTIONS:
Other: Braquial ecography — At the moment of the ecography, the clinician evaluates the endothelial responses via applying braquial ischemia and administering sublingual nitroglicerin spray to evaluate vasodilation.

SUMMARY:
The purpose of this study is to determine whether tocilizumab changes the cardiovascular risk factors on patients with arthritis rheumatoid.

Study hypothesis: the IL-6 contributes to increase the cardiovascular risk factors of patients with rheumatoid arthritis because it produces systemic effects as increasing weight and atherogenic body fat, changing energy homeostasis and inducing the adipokines production and the insulin resistence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and <70 years.
2. Diagnosis of active Rheumatoid Arthritis, moderate to severe (≥ 3.2 DAS28) of ≥ 6 months duration.
3. Patients with an inadequate clinical response to a stable dose of non-biological DMARDs or anti-TNF treatment for a period ≥ 8 weeks before treatment.
4. If patients are receiving oral corticosteroids, the dose should have been ≤ 10 mg predinosona and stable for at least one month before the start of treatment (day 1).
5. Patients who are able and wish to sign the informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Major surgery (including joints surgery) within eight weeks prior to the screening visit or major surgery scheduled for six months after first infusion.
2. Other Rheumatic autoimmune diseases, including systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis or systemic involvement secondary to AR (such as vasculitis, pulmonary fibrosis or Felty's syndrome). It's allowed the inclusion of patients with interstitial pulmonary fibrosis and be still able to tolerate treatment with MTX. Sjögren's syndrome with RA is not considered exclusion criterion.
3. Rheumatoid arthritis with Functional Class IV as defined in the RA Classification of the ACR (complete or significant disability of patients, confined to bed or to the wheelchair and without possibilities to take care themselves).
4. Prior or actual inflammatory joint disease different of RA (eg, gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease).

   Specific drug criteria
5. Treatment with any investigational agent in the four weeks before the screening visit (or time equivalent to five half-lives of the investigational drug, whichever is longer).
6. Immunization with a live vaccine / attenuated in the four weeks prior to the baseline visit.
7. Pretreatment with TCZ Laboratory Tests (at the screening visit)
8. Serum creatinine> 142 mmol / l (1.6 mg / dL) in women and> 168 mmol / l (1.9 mg / dl) in men and absence of active renal disease.
9. ALT (SGPT) and AST (SGOT)> 1.5 ULN (if the initial sample of ALT [SGPT] or AST [SGOT] gives a value> 1.5 times ULN, you can take and analyze a second sample during the selection period).
10. Platelet count <100 x 109 / l (100.000/mm3).
11. Hemoglobin <85 g / dl (<8.5 g / l, 5.3 mmol / l).
12. Leukocytes <1.0 x 109 / l (1000/mm3), ANC <0.5 x 109 / L (500/mm3).
13. RAL <0.5 x 109 / L (500/mm3).
14. Positivity for surface antigen of hepatitis B (HBsAg) and antibodies to hepatitis C.
15. Total bilirubin> ULN (if the initial sample of bilirubin> ULN, you can take and analyze a second sample during the selection period).
16. Triglycerides> 10 mmol / l (> 900 mg / dl) at the screening visit (non fasting).
17. Pregnant or lactating women.
18. not use of reliable means of contraception, such as a physical barrier (patient and partner), pill or contraceptive patch, spermicide and barrier or IUD.
19. Background of serious allergic or anaphylactic reactions to human monoclonal antibodies, humanized or murine.
20. RXT evidence of clinically significant abnormality.
21. Evidence of uncontrolled concomitant serious illness, cardiovascular, nervous system, lung (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), or gastrointestinal.
22. history of diverticulitis, diverticulosis in antibiotic treatment, the physician should consider the benefit-risk ratio.
23. Background of lower GI ulcer disease as the Crohn's disease, ulcerative colitis or other symptomatic conditions predisposed to perforations lower GI
24. Uncontrolled diseases such as asthma, psoriasis or inflammatory bowel disease,... treated normally with corticosteroids orally or parenterally.
25. Ongoing liver disease as determined by the principal investigator. (Patients with a history of elevated ALT (SGPT) will not be excluded)
26. Active infections or recurrent infections in the past by mycobacteria, fungus, virus or bacteria (for example: tuberculosis, atypical mycobacterial disease, clinically significant abnormalities in RXT, hepatitis B and C, herpes zoster), or any major episode infection that required hospitalization or IV antibiotic treatment in the 4 weeks preceding the screening visit or oral antibiotic in the 2 weeks prior to the screening visit.
27. Primary or secondary immunodeficiency.
28. Evidence of active malignancy diagnosed within 5 years before the inclusion(including solid tumors and hematological), or breast cancer diagnosed in the previous 5 years.
29. Active tuberculosis (TB) requiring treatment within 3 years above. Patients with a positive skin test tuberculin purified protein derivative (PPD) at the screening visit. Patients treated for tuberculosis no recurrence in the last three years will not be excluded.
30. HIV positive patients.
31. History of alcoholism, drug addiction or drug abuse in the six months before the screening visit.
32. Painful neuropathies or other conditions that may interfere with the pain assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Framingham Point Scores | Baseline and 52 weeks
  Proportion of changes in Framingham Point Scores

SECONDARY OUTCOMES:
Liver enzymes | Baseline, 12, 24 and 52 weeks
  Number of patients with liver enzymes elevated.
Lipoprotein levels | Baseline, 12, 24 and 52 weeks
  Number of patients with elevated lipoprotein levels
DAS28 score | Baseline and 52 week
  Variation in DAS28 score after tocilizumab
Number of patients with Adverse Drug Reactions | up to 52 weeks
  Number of patients with Adverse Drug Reactions as a measure of safety
Insulinemia | Baseline and 52 week
  Change in insulinemia 52 weeks later.

OTHER OUTCOMES:
Proportion of brachial artery vasodilation | Baseline, 24 and 52 weeks
  To evaluate the endothelial responses to ischemia and vasodilatation by ecography
cytokines, adipokines and adhesion molecules levels | Baseline and 52 week
  To evaluate changes in cytokines, adipokines and adhesion molecules

CONTACTS AND LOCATIONS:
Overall Officials: Federico Díaz González, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain